CLINICAL TRIAL: NCT04276870
Title: CD19-Directed Chimeric Antigen Receptor CD19 Redirected Autologous T Cells (CART19) for Orphan Indications of Pediatric B Cell Acute Lymphoblastic Leukemia (B ALL)
Brief Title: Orphan Indications for CD19 Redirected Autologous T Cells
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephan Grupp MD PhD (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, Stephan Grupp MD PhD, Director, Cancer Immunotherapy Program, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 834653, 19CT023, 19-016979
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-01

CONDITIONS: Pediatric and Young Adult Patientswith Hypodiploid or t(17;19) B-ALL; Infants With Very High Risk KMT2A B-ALL; Patients With Central Nervous System Relapse Who Did Not Receive Cranial Radiation or Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Subjects with hypodiploid B-ALL (Experimental)
  Interventions: Biological: Murine CART19
- Subjects with t(17;19) B-ALL (Experimental)
  Interventions: Biological: Murine CART19
- Infant subjects with very high risk KMT2A B-ALL (Experimental)
  Interventions: Biological: Murine CART19
- Subjects with central nervous system (CNS) relapse (Experimental): who did not receive cranial radiation (XRT) or bone marrow transplantation (BMT)
  Interventions: Biological: Murine CART19

INTERVENTIONS:
Biological: Murine CART19 — CART19 cells transduced with a lentiviral vector to express anti-CD19 scFv:41-BB:TCRζ, administered by IV injection with a planned dose of 5x106 CART19 cells/kg on day 0 with possible reinfusion/retreatment

SUMMARY:
This is an open-label, four-cohort, phase 2 study to determine the efficacy of CART19 in pediatric and young adult patientswith hypodiploid (Cohort A) or t(17;19) B-ALL (Cohort B), infants with very high risk KMT2A B-ALL (Cohort C), and in patients with central nervous system (CNS) relapse who did not receive cranial radiation (XRT) or bone marrow transplantation (BMT) (Cohort D).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form must be obtained prior to any study procedure.
2. Male and female patients with documented CD19+ B-ALL

   a.Cohort A & B: Patients, regardless their response to initial or relapsed B ALL therapy, with the following characteristics: i.Cohort A: Subjects with confirmation of a hypodiploid karyotype (chromosome number fewer than 45) ii.Cohort B: Subjects with cytogenetic confirmation of the chromosomal translocation t(17;19) (Cohort B) b.Cohort C: Infants w/ newly diagnosed KMT2A rearranged B-ALL classified as very high risk by the following criteria: i.Age < 3 months at diagnosis ii.Age < 6 months and WBC > 300,000x109/L at diagnosis or a poor prednisone response in induction iii.MRD positive > 0.01 (or PCR > 104) after 2 courses of standard infant ALL therapy.

   c.Cohort D: Subjects in a first or greater CNS relapse, prior to therapy with cranial XRT or HSCT for the current relapse
3. Documentation of CD19 tumor expression in bone marrow, peripheral blood, CSF, or tumor tissue.
4. Age 0 to 29 years
5. Adequate organ function defined as:

   1. A serum creatinine based on age/gender as follows:

      Maximum Serum Creatinine (mg/dL) Age Male Female 0 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1.0 1.0 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

      ≥ 16 years 1.7 1.4
   2. Adequate liver function:

   i.ALT≤ 5 x ULN; ALT ii.Total bilirubin ≤ 3 x ULN iii.ALT and/or bilirubin results that exceed this range are acceptable if, in the opinion of the physician-investigator (or as confirmed by liver biopsy), the abnormalities are directly related to ALL infiltration of the liver.

   c.Must have a minimum level of pulmonary reserve defined as ≤ Grade 1 dyspnea and < Grade 3 hypoxia; DLCO ≥ 40% (corrected for anemia) if PFTs are clinically appropriate as determined by the physician-investigator.

   d.Left Ventricular Shortening Fraction (LVSF) ≥ 28%, or Left Ventricular Ejection Fraction (LVEF) ≥ 45% by echocardiogram. In cases where quanitative assessment of LVSF/LVEF is not possible, a statement by the cardiologist that the ECHO shows qualititatively normal ventricular function wll suffice.
6. Adequate performance status defined as Lansky or Karnofsky score ≥ 50
7. Subjects of reproductive potential must agree to use acceptable birth control methods

Exclusion Criteria:

1. For subjects with a CNS relapse, prior cranial XRT or BMT for the current relapse is an exclusion.
2. Active hepatitis B or active hepatitis C.
3. HIV Infection.
4. Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy.
5. Concurrent use of systemic steroids at the time of cell infusion or cell collection, or a condition, in the treating physician's opinion, that is likely to require steroid therapy during collection or after infusion. Steroids for disease treatment at times other than cell collection or at the time of infusion are permitted. Use of physiologic replacement hydrocortisone or inhaled steroids is permitted as well.
6. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity.
7. Pregnant or nursing (lactating) women.
8. Uncontrolled active infection.

Ages: 0 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2028-03-10 (Estimated); Study Completion 2037-03-10 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | One year
  1 year event-free survival (EFS), where events include no response, relapse, death due to any cause

SECONDARY OUTCOMES:
EFS Rate 1 | One year
  Modified EFS rate in CNS relapse patients, using a definition of events that includes no response, relapse, death, need for XRT or need for BMT
To further evaluate the safety of CART19 in the target patient populations | One year
  Frequency and severity of adverse events
EFS rate 2 | One year
  Modified EFS rate in patients with early CNS relapsed B-ALL (CR1 <18 months) and those with late CNS relapsed B-ALL (CR1 >18 months) using a definition of events that includes no response, relapse, death, need for XRT or need for BMT
MRD conversion | One year
  Rate of MRD conversion to less than 0.01% (in patients with MRD) 28 days after CART19 therapy in patients with t(17;19) B-ALL, hypodiploid B-ALL, and very high risk infant B-ALL
Relapse Free survival 1 | One year
  Relapse-free survival (RFS) at one year in patients with hypodiploid B-ALL, patients with t(17;19) B-ALL, and very high risk infant B-ALL regardless of their initial response to B-ALL therapy and in patients with CNS relapse who did not receive cranial XRT or BMT after CART19 and who achieved a complete remission following CART19 therapy.
Relapse Free survival 2 | One year
  RFS at one year in patients with hypodiploid B-ALL who were MRD negative at end of induction and those who were MRD positive at end of induction during upfront therapy
Relapse Free survival 3 | One year
  RFS at one year in patients with t(17;19) B-ALL who were MRD negative at end of induction and those who were MRD positive at end of induction during upfront therapy
Relapse Free survival 4 | One year
  RFS at one year in very high risk infants with KMT2A rearrangement who were MRD negative at end of induction and those who were MRD positive at end of induction.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Grupp, MD, PhD, Study Director — Children's Hospital of Philadelphia; Amanda DiNofia, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No